CLINICAL TRIAL: NCT00903643
Title: Sensory Processing in Subjects With Painful Bladder Syndrome
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Washington University Early Recognition Center (Other)
Responsible Party: Sponsor
Other Study IDs: F08047007
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Painful Bladder Syndrome
Keywords: Painful Bladder Syndrome; Urinary Bladder
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy subjects
  Interventions: Other: Physical examination
- PBS subjects
  Interventions: Other: Physical examination

INTERVENTIONS:
Other: Physical examination — Physical examination and multiple questionnaires will be administered

SUMMARY:
The purpose of this study is to determine if clinically relevant subsets exist in patients meeting the diagnosis of Painful Bladder Syndrome (PBS). Subsets suggest differential responses to treatments and if verified, this will be important for the stratification of patients in clinical studies related to PBS.

DETAILED DESCRIPTION:
Patients with the diagnosis of painful bladder syndrome (PBS) constitute two or more phenotypes that are distinguished by differential neurophysiological processing of sensory information. Further, these differing phenotypes can be predicted by the presence or absence of the co-morbidity fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* NIDDK criteria for Painful Bladder Syndrome
* Age 19 years or older
* Must be able to read and speak English since testing materials are validated in English

Exclusion Criteria:

* PBS subjects must be independent of co-existing pain disorders or use of medications
* Uncontrolled hypertension or significant cardiopulmonary disease
* No chronic daily pain
* Older than 75 years of age

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with condition will be from Kirklin Clinic Urology Clinic and the Highlands Pain Treatment Clinic. Healthy subjects will be recruited via advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
This study proposes to examine the sensations that are produced by warming the skin, poking the skin, pressure on muscles and by applying a blood pressure cuff. | One and half to two hours.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Ness, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Kirklin Clinic Urology Clinic, Birmingham, Alabama, United States